CLINICAL TRIAL: NCT04580056
Title: Oocyte Recipients Before Embryo Transfer Randomization: Hysteroscopy With Fundus Uterus Scratching VS Hysteroscopy Without Fundus Uterus Scratching
Brief Title: Hysteroscopy With Fundus Uterus Scratching Incision VS Office Hysteroscopy Before ET With Donor Eggs
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assisting Nature (Other)
Collaborators: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Papanikolaou Evaggelos, Prof Dr Papanikolaou G. Evangelos, Assisting Nature
Other Study IDs: Uterus Incision- Don
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Hysteroscopy, Oocyte Recipients
Keywords: Hysteroscopy; Fundus Endometrial Incision; Oocyte acceptors; pregnancy outcome; uterine scratching

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Incision Group: Women following IVF treatment with donor oocytes who underwent during hysteroscopy fundus endometrial scratching by incision, before embryo transfer.
  Interventions: Procedure: Uterine fundus endometrial incision during hysteroscopy
- No incision Group: Women following IVF treatment with donor oocytes who underwent office hysteroscopy without fundus endometrial scratching by incision, before embryo transfer.

INTERVENTIONS:
Procedure: Uterine fundus endometrial incision during hysteroscopy — Uterine fundus endometrial scratching during hysteroscopy by incision
  Groups: Incision Group

SUMMARY:
A prospective randomised control trial of the impact of the fundus edometrial incision during hysteroscopy in oocyte recipients.

DETAILED DESCRIPTION:
A prospective randomised control trial of the impact of the fundus edometrial incision during hysteroscopy in women without intrauterine pathology which is likely to have an adverse effect on reproductive outcomes. The study populations will be constituted by oocyte recipients.

Study group: Hysteroscopy with fundus endometrial incision Control group: Office Hysteroscopy without any endometrial injury

ELIGIBILITY:
Inclusion Criteria:

* oocyte acceptors
* age 30-50
* embryo transfer with Hormone Replacement Therapy
* embryo transfer within 6 months of hysteroscopy

Exclusion Criteria:

* previous uterine pathology
* sperm sample <1mil/ml
* leiomyoma
* septate uterus

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women 30-50 years old with infertility undergoing IVF treatment with donor oocytes. 1-2 blastocysts are transferred per cycle with endometrium preparation with Hormone Replacement Therapy.The study population has underwent hysteroscopy with fundus endometrial incision before the embryo transfer.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Implantation Rate | 6 weeks to 42 weeks after embryo transfer]
  Implantation rate
Delivery Rate | 6 weeks to 42 weeks after embryo transfer]
  Delivery Rate

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Papanikolaou, PhD, Principal Investigator — Assisting Nature, 3rd Department of Obstetrics and Gynaecology, Aristotle University of Thessaloniki
Locations (1):
- Assisting Nature, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peitsidis N, Tsakiridis I, Najdecki R, Michos G, Kalogiannidis I, Athanasiadis A, Papanikolaou E. Hysteroscopic Endometrial Fundal Incision versus Hysteroscopy Only in Oocyte Recipients: A Randomized Controlled Trial Assessing The Reproductive Outcomes. Int J Fertil Steril. 2024 Jul 13;18(Suppl 1):3-9. doi: 10.22074/ijfs.2024.2009369.1523. PMID 39033364